CLINICAL TRIAL: NCT04112732
Title: Improving Everyday Functioning in Adults Aged 70 and Over Using a Multivitamin Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Vitabiotics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17016
Record Dates: First submitted 2019-08-30; First posted 2019-10-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2022-12

CONDITIONS: Aging; Stress
Keywords: Multivitamin; Aging; Stress; Everyday Function; Well-Being
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multivitamin (Experimental): 1 multivitamin tablet administered by mouth daily for 12 weeks, to be taken with main meal.
  Interventions: Dietary Supplement: Multivitamin
- Placebo (Placebo Comparator): 1 placebo tablet administered by mouth daily for 12 weeks, to be taken with main meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin — Multivitamin
  Arms: Multivitamin
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Investigation of the chronic effect of 12 week multivitamin supplementation on markers of everyday function in adults aged 70 and over.

DETAILED DESCRIPTION:
Everyday functioning relates to how well an individual can function independently in day-to-day life. As a person ages, there are various changes which occur in the body, which can lead to a decline in everyday functioning. There is a loss of bone density, the immune system naturally declines which can lead to a susceptibility to autoimmune diseases, infection and cardiovascular disease. Many older adults report feeling socially isolated and lonely, which can also lead to poor mood and negative health outcomes. Due to advancements in society, there has been an increase in older adult informal caregivers, which is a form of chronic stress associated with a range of negative outcomes and declines in functioning.

Nutritional supplementation may have the potential to improve everyday functioning in older adults, which may have declined through ageing alone or ageing alongside chronic stress from being a caregiver. Research had shown multivitamin supplementation to have positive cognitive, mood, mobility and health effects. As well as improving general day-to-day well-being and functioning, and may have the ability to reduce feeling of stress.

The current study will investigate the effects of a multivitamin supplement following daily intake for 12 weeks on a range of everyday functioning outcomes in adults aged 70 and over. The outcome measures include; well being, cardiovascular reactivity, immune response, stress, self-reported health, daily functioning behaviours, mobility, mood, cognitive function, sleep quality and loneliness.

Amendment to protocol:

The recent Covid-19 restrictions have led to changes to the original protocol. Specifically, a group of participants who completed their baseline assessment as per the outlined protocol could not complete the final testing visit as initially planned because of the imposed lockdown For these participants, all follow-up questionnaire-based assessments have been conducted online from their home.

These necessary changes to the method of data collection will be a confounding factor in this group, which would not be comparable to the main dataset. Therefore, the decision has been made to un-blind the researcher to this group of participants' treatment (11 who completed in full prior and 34 who completed testing visit 2 online).

This will allow the main outcome measures to be compared in this unique group of participants', as well as comparisons between outcome measures in those who completed pre and during lockdown.

ELIGIBILITY:
Inclusion Criteria

* Aged over 70
* Both caregivers and non caregivers will be recrtuied

Exclusion Criteria

* Allergy to soya
* Participants must not be currently taking the investigational product (or another equivalent multivitamin); any participants who report multivitamin use must be willing to have a washout for 4 weeks before participating (if not willing to do this they will be excluded)
* If a participant has epilepsy, a thyroid disorder, haemochromatosis or suffers from food allergies they must consult their doctor/pharmacist before taking part

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-11-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Well-Being (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  An overall outcome measure which is a composite measure made up of four personal well-being questions used in the Measuring National Well-being programme plus one additional question.
  These five questions are:
  1. Overall, how satisfied are you with your life nowadays?
  2. Overall, to what extent do you feel the things you do in your life are worthwhile?
  3. Overall, how happy did you feel yesterday?
  4. Overall, how anxious did you feel yesterday?
  5. Overall, how well did you feel yesterday?

SECONDARY OUTCOMES:
Cardiovascular reactivity- Blood pressure (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Systolic and Diastolic blood pressure measured via Portapres a non-invasive, continuous beat-to-beat blood pressure monitoring system.
Cardiovascular reactivity- Heart rate (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Beats per minute, measured via Portapres a non-invasive, continuous beat-to-beat blood pressure monitoring system.
Immune/inflammatory response (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  C-Reactive Protein (CRP)
Immune/inflammatory response(change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Secretory Immunoglobulin-A (s-IgA)
Self-Reported Stress (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  The Kingston Caregiver Stress Scale.This tool is designed to assess levels of perceived stress associated with caregiving in informal carers. The scale comprises three sections that assess levels of stress in relation to care-related feelings; family matters; and financial stresses. Higher scores indicate higher levels of stress
Self-Reported Stress (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  The Perceived Stress Scale (PSS), The PSS is a 10-item scale which measures the extent to which participants perceive their lives to be overwhelming, uncontrollable and unpredictable.Scale responses range from 0 (never) to 4 (very often) and items are summed to yield a total score. Higher scores indicate greater perceived levels of stress, experienced over the previous month
General health(change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Cohen Hoberman Inventory of Physical Symptoms.The CHIPS was designed as a measure of perceived burden due to the experience of a range of physical symptoms. The scale comprises a list of 33 common everyday symptoms (e.g. 'acne', 'diarrhoea', 'heart pounding or racing') and asks respondents 'how much that problem has bothered or distressed you during the past two weeks including today'. Items are scored for 1-5, then summed across all items. Higher scores indicate worse health
General health (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  SF-20. The survey measures health across 6 domains: physical functioning (6 questions), role functioning (2 questions), social functioning (1 question), mental health (5 questions), health perceptions (5 questions), and pain (1 question).Scores across each of these domains are reported on a 0% to 100% scale, with 0% representing the worst possible score in that domain and 100% the best possible score. Raw scores are transformed to fit the 0% to 100% interval as described in the original publication (note that for question #1 on general health, an initial transformation is performed as follows: 1 = 5, 2 = 4.36, 3 = 3.43, 4 = 1.99, 5 = 1). Reversal of scoring is completed as necessary such that the highest score always represents the best possible score. The exception to this scoring pattern is the pain score, for which 0% represents the best possible score and 100% the worst possible score,
Daily functioning and care behaviours (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Instrumental Activities of Daily Living Scale. is an appropriate instrument to assess independent living skills.There are eight domains of function measured with the Lawton IADL scale.
  Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded.
  Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
Mood trait measures (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Hospital Anxiety and Depression Scale, this is a 14 item scales, with scale responsed rangin from 0 to 5. Scores are summed to produce separate scores for anxiety and depression. Higher scores indicate more frequent feelings of anxiety and depressive symptoms. Scores between 0 and 7 are considered normal. Scores between 8 and 10 are indicative of borderline mood disorder and scores > 11 indicates probable mood disorder
Mood trait measures (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Profile of Moods States (POMS). This comprises 37 items with response ranging from 'not at all' to 'extremely'. Scores from the POMS-SF are used to derive a total score for 'mood disturbance', as well as subscores for the domains of 'tension', 'depressed', 'anger', 'vigour', 'fatigue' and 'concentration'. A total score disturbance score can also be calculated by adding the scores from the first five of these global scores and subtracting 'vigour
Acute measures of subjective state in responses to a stressor (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  State-Trait Anxiety Inventory (STAI) The STAI is a widely used instrument consisting of two subscales assessing 'State' and 'Trait' anxiety respectively. Each subscale contains 20 statements (e.g. 'I am calm') each with a 4-point Likert scale, giving a range of potential scores from 20 to 80. Participants rate how much they feel like each statement at the time of making the response (State subscale), and how much they generally feel like each statement (Trait subscale). Higher scores indicate greater anxiety.
Acute measures of subjective state in responses to a stressor (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  NASA-Task Load Index. The NASA-TLX comprises a set of six scales anchored with 'Low' and 'High' at the extreme points. Three of the scales reflect the demand placed upon the respondent by the task (Mental Demand, Physical Demand, Temporal Demand), whereas three reflect the interaction between the respondent and the task (Effort, Perceived Performance, Frustration).
Cognitive function (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Task performance on the Multi-Tasking Framework (MTF),
Cognitive function (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Prospective and Retrospective memory Questionnaire, The PRMQ is a 16 item scale that quantifies memory failures for everyday tasks over two subscales: prospective memory (e.g., do you forget appointments if you are not prompted by someone else or by a reminder such as a calendar or diary?) and retrospective memory (e.g., do you fail to do something you were supposed to do a few minutes later even though it's there in front of you, like take a pill or turn off the kettle?). Scale responses range from 1 (never) to 5 (very often), and higher scores indicate poorer everyday memory.
Cognitive function (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  A covert measure of prospective memory, whereby participants will be asked to remember to return a reminder slip with their 'participant number' written on, which will be posted out before testing visits.
Sleep quality (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Pittsburgh Sleep Quality Index. The PSQI assesses seven factors - subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction - via questions regarding sleep timings and zero to three-point scales in which participants rate whether they have experienced a number of issues (e.g. 'During the past week, how often have you had trouble sleeping because you have had bad dreams?') from 'not during the past week' to '3 or more times in the past week'. A global sleep score is created by totalling the seven subfactor scores, with higher scores indicating poorer sleep quality.
Mobility (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Yale Physical Activity Scale, The YPAS is an interviewer-administered questionnaire developed to assess physical activity in older adults. The YPAS is divided into two sections: in the first section, there is a comprehensive physical work, exercise, and recreational activities checklist to assess time spent in these types of activities during a typical week in the past month. The second section contains questions to quickly assess an individual's participation in five activity dimensions: vigorous activity, leisurely walking, moving on feet, standing, and sitting. Responses on the YPAS allow eight summary indices to be calculated: total time spent per week in all physical activities, weekly energy expenditure in kcal per week, five individual indices for the activity dimensions, and an activity dimension summary index
Mobility (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Falls Efficacy Scale, measures of "fear of falling" or, more properly, "concerns about falling.To calculate the FES-I score when all items are completed, simply add the scores for each item together to give a total that ranges from a minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Mobility(change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Timed up and Go Test, length of time in seconds it takes participants to stand form a chair, walk 3 metres, turn around and sit back down in chair.
Mobility (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Grip Strength. 3 trials on non dominant hand. Measured in kg.
Mobility(change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Balance tests. Measured to see if participants can hold 3 stances for 10s. If they can they are awarded 1 point, if not 0 points.
Social network size (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Lubben Social Network Scale, This measure uses 6 questions: 3 key questions evaluate the size of 3 different aspects of social network that are attributable to family ties and a parallel set attributable to friendship ties. Each LSNS-6 question is scored on a 0 to 5 scale. The total score is an equally weighted sum of these 6 questions, with scores ranging from 0 to 30.
Social network size (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  Convoy Method. • Respondents are presented with a set of three concentric circles, with the word 'You' contained within a smaller circle in the middle. Respondents are asked to think about "people who are important in your life right now, but who are not equally close". Respondents are then asked to think about "people to whom you feel so close it is hard to imagine life without them"; these people are entered into the innermost circle. For the next circle respondents are asked to consider "people to whom you may not feel quite that close but who are still very important to you". Finally, in the outer circle respondents are asked to place "People whom you haven't already mentioned but who are close enough and important enough in your life that they are part of your personal network". The numbers of people within each network are counted and can be used to represent support networks in each of the categories and / or summed to produce an index of total social network size
Loneliness (change from baseline) | Measured at baseline and then following chronic (12 weeks) treatment
  The De Jong Gierveld Loneliness Scale,This tool can be used to provide a single index of loneliness in addition to indices of 'Emotional Loneliness' and 'Social Loneliness' . To score the answers to the scale, the neutral and positive answers are scored as "1" on the negatively worded questions and On the positively worded items, the neutral and negative answers are scored as "1"
Nutrition Status | Measured at baseline and then following chronic (12 weeks) treatment
  Blood biomarkers taken to assess impact of nutritional status, this will measure vitmain B12, ferritin and folate.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No